CLINICAL TRIAL: NCT05990699
Title: Effect of Mindfulness-Based Relapse Prevention Program on Readiness for Change and Self-efficacy Among Clients With Substance Use Disorders: A Randomized Control Trial
Brief Title: Effect of Mindfulness-Based Relapse Prevention Program on Readiness for Change and Self-efficacy Among Clients With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed El-Ashry, Lecturer at psychiatric and mental health nursing, faculty of nursing, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00013620/7/2023
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Substance Use Disorders
Keywords: Mindfulness; Relapse Prevention; Readiness for Change; Self-efficacy; substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): patients will under routine hospital care as well as MBRP. This program consists of eight sessions spanning across four weeks, each focusing on specific techniques and skills to aid in substance use disorder treatment. The first session emphasizes the correlation between the "unconscious pilot" and substance use, incorporating a "corporeal examination" technique to promote intentional concentration. The second session focuses on mindfulness to identify stimuli and observe accompanying sentiments, thoughts, and feelings. The third session introduces the "ABSTEMIOUS space" technique, urging patients to pause, observe their experiences, concentrate on breathing, broaden cognizance, and choose judicious responses in trying or hazardous situations. The remaining sessions address coping mechanisms for relapse risks, taking pragmatic action in high-risk situations, integrating healthy activities into life, and sustaining mindfulness practice through the development of a support network.
  Interventions: Behavioral: Mindfulness-Based Relapse Prevention program
- control group (No Intervention): patients with substance use disorder who will be under routine hospital care.

INTERVENTIONS:
Behavioral: Mindfulness-Based Relapse Prevention program — This program consists of eight sessions spanning across four weeks, each focusing on specific techniques and skills to aid in substance use disorder treatment. The first session emphasizes the correlation between the "unconscious pilot" and substance use, incorporating a "corporeal examination" technique to promote intentional concentration. The second session focuses on mindfulness to identify stimuli and observe accompanying sentiments, thoughts, and feelings. The third session introduces the "ABSTEMIOUS space" technique, urging patients to pause, observe their experiences, concentrate on breathing, broaden cognizance, and choose judicious responses in trying or hazardous situations. The remaining sessions address coping mechanisms for relapse risks, taking pragmatic action in high-risk situations, integrating healthy activities into life, and sustaining mindfulness practice through the development of a support network.
  Arms: Intervention group

SUMMARY:
The treatment process of substance addiction is applied principally by psychiatrists, psychologists, and psychiatric mental health nurses. In this respect, psychiatric mental health nurses have a crucial role to play. As they are the one who is in touch with the patients for 24 hours, psychiatric nurses can enhance the treatment process a lot through the application of a mindfulness-based relapse prevention program.

As drug abuse is such a devastating affliction, further knowledge about specific traits that may increase the chances of a successful recovery would be greatly beneficial to enhance treatment and decrease relapse rate. Accordingly, this study will be conducted to determine the effect of mindfulness-based relapse prevention program on readiness for change, and efficacy among clients with substance use disorder.

AIMS OF THE STUDY

The aim of this study is to:

Examine the effect of the Mindfulness-Based Relapse Prevention Program on readiness for change and self-efficacy among clients with substance use disorder during the rehabilitation phase.

RESEARCH HYPOTHESIS Clients with substance use disorder who attend Mindfulness-Based Relapse Prevention program sessions exhibit higher levels of readiness for change and self-efficacy compared to those who receive conventional hospital treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write.
* Able to communicate and willing to participate in the study.
* Male patients only Exclusion Criteria
* Patients who are only alcoholics will be excluded.
* Diagnosed with SUDs with mental illness comorbidity.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male patients only to decrease confounding factors
Enrollment: 100 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Five Factors Mindfulness Questionnaire (FFMQ) | 5 weeks
  This scale was developed by Baer et al (2006) to measure elements of mindfulness (104). It is composed of 39-items, which are rated on a five point likert scale. The responses ranging from 1 (never or very rarely true) to 5 (very often or always true). The scale is divided into five subscales which are observing (notice or attend to internal and external phenomena), describing (label observed phenomena such as thoughts and emotions), acting with awareness (engage with full awareness in current experience or activity), non-judging of inner experience (nonjudgmental awareness of current experience without evaluation) and non reactivity to inner experience (notice internal phenomena without reacting).
  . Higher scores of the subscales represent greater observing, describing, awareness, non- judgment and non reactivity.
The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) | 5 weeks
  This scale was developed by Miller and Tonigan (1996) to assess readiness for change in alcohol and substance abuse clients (version 8D) (Miller & Tonigan., 1996). It is composed of 19-items, which are rated on a five-point Likert scale. The responses ranged from 1 (No, strongly disagree) to 5 (Yes, strongly agree). The scale includes statements belonging to three factors of readiness for change which are Recognition, Ambivalence, and Taking Steps. The nineteen items have a total score ranging from 19 to 95, with higher scores indicating higher levels of recognition, ambivalence and taking steps.
Drug abstinence Self-Efficacy Scale (DASE) | 5 weeks
  DASE scale is a modified version of Alcohol Abstinence Self- Efficacy scale. It was modified by Hiller et al (2000). It is composed of 20-items, which are rated on a five-point Likert scale ranging from 1 (not at all) to 5 (extremely). The scale encompasses four subscales, five items each that examine cues related to: negative affect, social interactions & positive states, physical & other concerns and finally Cravings & urges. For each item, respondents are requested to respond to how "tempted" they would be to use drugs in each situation. The same 20 items are presented to the subjects for a second time but this time they are requested to indicate how "confident" they are that they would not use drugs in that situation (abstinence self-efficacy). The twenty items are summed to obtain a total score that ranges from 20 to 100 with higher scores reflecting greater self-efficacy for each temptation and confidence separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bowen S, Chawla N, Collins SE, Witkiewitz K, Hsu S, Grow J, Clifasefi S, Garner M, Douglass A, Larimer ME, Marlatt A. Mindfulness-based relapse prevention for substance use disorders: a pilot efficacy trial. Subst Abus. 2009 Oct-Dec;30(4):295-305. doi: 10.1080/08897070903250084. PMID 19904665